CLINICAL TRIAL: NCT01339026
Title: Evaluating the Benefit of Additional Platelet Inhibition in Acute Coronary Syndrome Patients With High Platelet Reactivity Undergoing PCI
Brief Title: Evaluating Additional Platelet Inhibition in Patients With High Platelet Reactivity Undergoing Percutaneous Coronary Intervention
Acronym: APACS-HPR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in guidelines favouring newer antiplatelet drugs in ACS
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-020219-35
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Cardiovascular Disease; Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Platelet reactivity; Clopidogrel; Percutaneous coronary intervention
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator): Day 1 loading 60mg Day 2 to 7 10mg o.d. Day 8 to 30 days 10mg od
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Day 1 Loading 600mg Day 2 to 7 day: 150mg o.d. Day 8 to 30 days: 75mg o.d.
  Interventions: Drug: Plavix

INTERVENTIONS:
Drug: Prasugrel — Day 1 loading 60mg Day 2 to 7 10mg o.d. Day 8 to 30 days 10mg od
  Other Names: Efient
  Arms: Prasugrel
Drug: Plavix — Clopidogrel (Plavix) Day 1 Loading 600mg Day 2 to 7 day: 150mg o.d. Day 8 to 30 days: 75mg o.d.
  Other Names: Clopidogrel
  Arms: Clopidogrel

SUMMARY:
Patients admitted to hospital with chest pain due to reduced blood flow to heart muscle (diagnosis Acute Coronary Syndrome) can be treated with medication and an angioplasty ± stent procedure, which restores blood flow to the heart. Antiplatelet drugs (Aspirin and Clopidogrel) are blood thinning treatments and research has reported they reduce heart attacks, death and stroke. The investigators know some patients do not respond fully to Clopidogrel but currently patients are not tested for this.

The investigators wish to perform a trial to identify those patients who do not respond fully to Clopidogrel and randomise them to either Prasugrel (newer drug) or a higher dose of Clopidogrel.

Patients admitted to the hospitals (2 in the UK and 1 in Germany) will be asked for their consent to participate. A blood sample is tested for platelet activity.

1. Low platelet activity result means patient has responded well to Clopidogrel and will continue on the routine dose. They will be entered into an observational registry. Data will be collected of routine blood tests and investigations, medication and procedures. Their GP will be contacted at about 30 days to see if they are alive.
2. High platelet activity results means patient has not responded fully to Clopidogrel. These patients will be randomly allocated to a higher dose of Clopidogrel or new drug Prasugrel. Data will be collected of routine blood tests and investigations, medication and procedures. A hospital visit at 30±5 days is required to assess how patients are doing, medications and occurrence of any events.

DETAILED DESCRIPTION:
STUDY DESCRIPTION This is a multinational, randomised open label study comparing Prasugrel versus Clopidogrel in ACS patients who have high platelet reactivity managed with an early invasive strategy (PCI as early as possible and no later than 72 hours from admission).

Patients identified with low platelet reactivity indicating a good response to Clopidogrel will be entered into an observational Registry.

Sites There will be three participating hospitals, two in the UK and one in Germany.

Screening All patients admitted to the hospital with suspected ACS requiring early PCI (within 3 days of admission) will be screened for entry into the trial.

The investigator and/or his/her designee will explain the study requirements and procedures and obtain consent before any study procedures are performed.

We estimate approximately 500 patients will be screened. From these a total of 140 patients will be randomised, the remaining screened patients will be entered into the registry. There will be competitive recruitment and each site is expected to randomise about 40 to 50 patients each. We estimate 7 to 8 patients randomised per month over a period of 18 months.

Routine blood tests and investigations will be carried out according to local management strategies. The angiogram and PCI procedure are part of the routine management for this patient and will be performed according to local policies and procedures.

A research blood sample will be required to determine platelet activity which has to be taken > 2hours from the standard Clopidogrel pre-PCI loading. For most patients this will be taken in the catheter laboratory around the PCI procedure. In a few patients who are loaded with Clopidogrel close to the PCI procedure the blood samples may be taken in the ward or recovery area. Depending on the platelet activity results patients will be either entered into the registry or randomly allocated to either Clopidogrel or Prasugrel.

1. Patients who are good responders to Clopidogrel (platelet reactivity <400 AUC min) will be entered into the registry.
2. Patients who are poor responders to Clopidogrel (platelet reactivity > 400AUC min) will be randomised.

REGISTRY PATIENTS Patients will continue on the standard treatment of Clopidogrel. Data will be collected of routine blood tests and investigations, medication and procedures. Additional blood samples will be taken (if patient consents) for the biomarker and genetic sub-studies. Their GP will be contacted at 30±5 days to see if they are alive.

RANDOMISED PATIENTS Randomisation Investigators will access an automated telephone or automated web service. Investigators will have to confirm patient fulfils the eligibility criteria and that consent has been obtained.

Randomised Treatment Randomised patients will be allocated to receive either open label Clopidogrel (Plavix) or Prasugrel (Efient).

Group 1: Clopidogrel (Plavix)

* Day 1 Loading 600mg
* Day 2 to 7 day: 150mg o.d.
* Day 8 to 30±5 days: 75mg o.d.

Group 2: Prasugrel (Efient)

* Day 1 loading 60mg
* Day 2 to 7 10mg o.d.
* Day 8 to 30±5 days 10mg od

Drug Supply and Storage Prasugrel, a commercially available product, will be supplied by Eli Lilly which holds the manufacturing license to produce Prasugrel. Clopidogrel (Plavix) will be purchased by the hospital Pharmacy through normal purchasing arrangements. All study drugs should be stored in an appropriate locked room, under the control of the Hospital Pharmacist or the Investigator, in the conditions described in the package insert.

Hospital Admission to Discharge

* Patients will be followed until they are discharged home.
* Blood samples taken for platelet activity at 1, 4 and 24 hours, and pre-discharge.
* Blood sample for the biomarker substudy will be taken pre-PCI procedure at 24 hours and at discharge.
* Blood sample for the genetic substudy will be taken at baseline or if not possible pre-discharge.
* Patients will have instructions on how to contact the research team if they have any questions or concerns.

One Month Follow UP RCT Patients in the RCT will be required to attend the hospital for a follow up visit at 30±5 days from date of randomisation. Patients will be assessed by the investigator or his/her designee for heart rate and blood pressure, medication tolerance and compliance, occurrence of adverse events and clinical endpoints, blood sample for platelet activity. At this time the investigator will discuss with the patient their treatment options after this period.

Sub-studies There are two sub-studies proposed (i) biomarker and (ii) genetic. Blood samples will be taken and stored locally before shipment to a core lab in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. ACS patients with intent for PCI <72 hours from admission.
2. Prior clopidogrel loading within 24h before planned PCI or chronic (>24 hours) treatment with clopidogrel
3. High platelet reactivity (HPR) PA > 400 AU min by multiplate analyser ("poor responders")
4. Initial platelet function sample at least 2 hours after pre PCI loading dose
5. Consent

Exclusion Criteria:

1. Patients <18 years and >75 years
2. Body weight <60kg
3. Pretreatment with prasugrel within 7 days of randomisation
4. History of stroke or transient ischaemic attack
5. Patients with increased bleeding risk e.g.

   * recent major trauma or surgery
   * gastrointestinal bleeding or active peptic ulceration
   * Platelet count <100,000 / mm3 at the time of screening
   * Internationally Normalized Ratio (INR)> 1.5 at the time of screening
6. Hb<10g/dL
7. Intracranial neoplasm, arteriovenous malformation or aneurysm.
8. Severe hepatic impairment (Child Pugh class C)
9. Intention to use the following medications

   * oral anticoagulation
   * other antiplatelet therapy (including GPIIb/IIIa inhibitors) besides aspirin
   * nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors
10. Female patients who are pregnant, planning pregnancy, not using reliable contraception or who are breastfeeding
11. Known allergy, hypersensitivity or other contraindications to prasugrel or clopidogrel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity | 4 hours post loading dose
  The primary endpoint will compare the proportion of patients with improved platelet response (i.e. decreased platelet reactivity under the cut-off value of 400 Au.min) in the prasugrel re-loading arm compared to the clopidogrel re-loading arm at 4 hours after randomization in patients with initial high platelet reactivity

SECONDARY OUTCOMES:
Platelet reactivity in response to randomised study drug | 7 days/hospital discharge and 30 days
  To compare the proportion of patients with improved platelet response between the treatment arms at hospital discharge/7 days and at 30 days.
Extent of myocardial damage | 24 hours
  To compare the AUC for CK and troponin at 24 hours between the treatment arms
MACE | 30 days
  To compare the rates major adverse events (death, myocardial infarction, stroke, repeated revascularization) at 30 days between the treatment arms
Bleed | 30 days
  To compare the rate of major bleedings at 30 days between the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Miles Dalby, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Tobias Geisler, MD, Principal Investigator — University Hospital Tuebingen; Azfar Zaman, MD, Principal Investigator — Freeman Hospital and University of Newcastle
Locations (1):
- Universitätsklinikum Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Geisler T, Booth J, Tavlaki E, Karathanos A, Muller K, Droppa M, Gawaz M, Yanez-Lopez M, Davidson SJ, Stables RH, Banya W, Zaman A, Flather M, Dalby M. High Platelet Reactivity in Patients with Acute Coronary Syndromes Undergoing Percutaneous Coronary Intervention: Randomised Controlled Trial Comparing Prasugrel and Clopidogrel. PLoS One. 2015 Aug 28;10(8):e0135037. doi: 10.1371/journal.pone.0135037. eCollection 2015. PMID 26317618